CLINICAL TRIAL: NCT00685425
Title: A Dose Response and PharmacoDynamic Study of Levalbuterol and Racemic Albuterol HFA MDI in Subjects Twelve Years of Age and Older With Asthma
Brief Title: Dose Response Study of Levalbuterol in the Prevention of Exercise Induced Bronchoconstriction Compared to Racemic Albuterol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 051-308
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma; Bronchoconstriction
Keywords: Asthma; Exercised induced bronchoconstriction
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects randomized to the levalbuterol arm will complete 1 of 6 possible randomization sequences containing (a) levalbuterol 45 µg (1 actuation of 45 µg); (b) levalbuterol 90 µg (2 actuation of 45 µg) and (c) levalbuterol 180 µg (4 actuations of 45 µg each). Subjects will receive treatment, according to the randomization sequence, followed by a 5±2 day washout.
  Interventions: Drug: Levalbuterol HFA MDI
- B (Active Comparator): Subjects randomized to racemic albuterol will complete 1 of 6 possible randomization sequences containing (a) racemic albuterol 90 µg (1 actuation of 90 µg); (b) racemic albuterol 180 µg (2 actuations of 90 µg) and (c) racemic albuterol 360 µg (4 actuations of 90 µg). Subjects will receive treatment, according to the randomization sequence, followed by a 5±2 day washout.
  Interventions: Drug: Racemic Albuterol

INTERVENTIONS:
Drug: Levalbuterol HFA MDI — 1. levalbuterol 45 µg (1 actuation of 45 µg); (b) levalbuterol 90 µg (2 actuation of 45 µg) and (c) levalbuterol 180 µg (4 actuations of 45 µg each).
  2. Arm #A
  3. Xopenex HFA MDI
  Arms: A
Drug: Racemic Albuterol — 1. racemic albuterol 90 µg (1 actuation of 90 µg); (b) racemic albuterol 180 µg (2 actuations of 90 µg) and (c) racemic albuterol 360 µg (4 actuations of 90 µg).
  2. Arm #B
  3. Proventil HFA MDI
  Arms: B

SUMMARY:
The purpose of this study is to investigate, using an exercise challenge approach, the dose response of levalbuterol HFA MDI in adolescent and adult subjects with asthma

DETAILED DESCRIPTION:
A randomized, modified-blind, active controlled, multicenter, parallel treatment, 3x3 dose level crossover study evaluating the dose response of levalbuterol in subjects 12 years of age and older with exercise induced bronchoconstriction. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, must be at least 12 years of age at the time of consent.
* Female subjects 12-60 years of age must have a negative serum pregnancy test.
* Women of child bearing potential must be using an acceptable method of birth control throughout the study.
* Subject must have a documented diagnosis of asthma for a minimum of 6 months prior to study start
* Subject must be in good health with the exception of their reversible airways disease and not suffering from any chronic condition that might affect their respiratory function.
* Subject must have a chest X-ray for the study or within 12 months prior to randomization.
* Subject must be able to complete the diary cards and medical event calendars reliably on a daily basis and understand dosing instructions. Any minor subject who is not able to do this must have a parent/legal guardian who can assist them during the study with these activities.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* Subject who has participated in an investigational drug study within 30 days of study start, or who is currently participating in another clinical trial.
* Subject whose schedule prevents him or her from starting study visits before 12 PM.
* Subject who is unwilling or physically unable to perform the exercise challenges as described in the protocol.
* Subject who has travel commitments during the study that would interfere with trial measurements or compliance or both.
* Subject who has a history of hospitalization for asthma within 4 weeks prior to study start, or who is scheduled for in-patient hospitalization, including elective surgery during the course of the trial.
* Subject with a known sensitivity to levalbuterol or racemic albuterol, or any of the excipients contained in any of these formulations.
* Subject using any prescription drug with which albuterol sulfate administration is contraindicated.
* Subject with currently diagnosed life-threatening asthma defined as a history of asthma episodes requiring intubation, associated with hypercapnia, respiratory arrest, or hypoxic seizures within 12 months prior to study start.
* Subject with a history of cancer (exception: basal cell carcinoma in remission).
* Subject with hyperthyroidism, diabetes, hypertension, cardiac diseases or seizure disorders that currently are not well controlled by medication or that may interfere with the successful completion of this protocol.
* Subject with a history of substance abuse or drug abuse within 12 months preceding study start. Urine drug test must be negative at study start.
* Subject with greater than 10 pack year history of cigarette smoking or use of any tobacco products within 6 months of study start.
* Subject with a documented history of bronchopulmonary aspergillosis or any form of allergic alveolitis.
* Subject who has suffered from a clinically significant upper or lower respiratory tract infection in the 3 weeks prior to study start.
* Subjects with unstable asthma; or who have had a change in asthma therapy; or a visit to the Emergency Department or hospital for worsening asthma within 4 weeks.
* Subject who is a staff member or relative of a staff member.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2002-10; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
FEV1 AUC 0-60 (% decrease from post-dose/pre-challenge FEV1) | Days -7, 0, 5, 10, 15

SECONDARY OUTCOMES:
Maximum percent decrease in FEV1 from visit post-dose/pre-challenge FEV1 | Days -7, 0, 5, 10, 15
Minimum percent change in FEV1 from visit pre-dose FEV1. | Days -7, 0, 5, 10, 15
time to recovery (min), Protected/Unprotected Subjects Counts | Days -7, 0, 5, 10, 15
FVC AUC 0-60 (% decrease from post-dose/pre-challenge FEV1). | Days -7, 0, 5, 10, 15
Maximum percent decrease in FVC from visit post-dose/pre-challenge FVC, | Days -7, 0, 5, 10, 15
Minimum percent change in FVC for pre-dose FVC, | Days -7, 0, 5, 10, 15
FEF25-75% AUC 0-60 (% decrease from post-dose/pre-challenge FEV1), | Days -7, 0, 5, 10, 15
Maximum percent decrease in FEF25-75% from visit post-dose/pre-challenge FEF25-75% | Days -7, 0, 5, 10, 15
Minimum percent change in FEF25%-75% from visit pre-dose FEF25-75%. | Days -7, 0, 5, 10, 15

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Los Angeles, California
  - Signal Hill, California
  - Denver, Colorado
  - Minneapolis, Minnesota
  - Burke, Virginia